CLINICAL TRIAL: NCT04162990
Title: Lifestyle Remodeling in Subjective Memory Complaint (SMC): Brain Imaging and Blood Biochemistry Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-06-002A
Record Dates: First submitted 2019-09-19; First posted 2019-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Subjective Memory Complaint
Keywords: Subjective Memory Complaint; Alzheimer's disease; mild cognitive impairment; Neuroinflammation; lifestyle
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neuroinflammatory Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle remodeling (Experimental)
  Interventions: Behavioral: Lifestyle remodeling Intervention
- Does Comparator: regular treatment (Active Comparator)
  Interventions: Behavioral: Does Comparator: regular treatment

INTERVENTIONS:
Behavioral: Lifestyle remodeling Intervention — Participants will be received 2 phases of intervention of lifestyle remodeling, 3 months for each phase, which contained cognitive stimulating activities and physical activities.
  Arms: Lifestyle remodeling
Behavioral: Does Comparator: regular treatment — Participants in this group would be treated as usual, which contained the healthy education.
  Arms: Does Comparator: regular treatment

SUMMARY:
The specific study aims:

1. To investigate whether the brain function is affected by the past life experiences, such as lifestyle and physiology-related factors in SMC.
2. To examine whether the lifestyle remodeling could improve SMC's cognitive function and modulate the reactivity of inflammatory factors, leading to significantly slow down the disease progression to MCI or dementia.
3. To investigate the lasting duration of the intervention.

DETAILED DESCRIPTION:
Although there is much evidence showing age-related reduction of cognitive function, many researchers point out a more optimistic viewpoint that aging is not a progressive loss. By remodeling the lifestyle, or/and monitoring the physical factors, the risk to develop dementia could be reduced. The above statements are mostly based on the epidemiological research, while it remains unclear how the aging modulates the brain changes. In previous study, the investigators have found that individuals with subjective memory complaint (SMC) showed altered brain changes in terms of resting-state connectivity when compared to those without SMC. The present study further aims to examine whether the brain function is affected by the past life experiences, such as lifestyle and physiology-related factors in SMC. More importantly, this study aims to clarify whether the lifestyle remodeling could improve SMC's cognitive function and modulate the reactivity of inflammatory factors, leading to significantly slow down the disease progression to MCI or dementia.

In summary, the present study aims to understand how the lifestyle remodeling affects SMC's brain function and biochemical indicators. Before and after the intervention, this study will use neuropsychological tests to assess all the aspects of cognitive functions, use Electroencephalogram to investigate the brain activation patterns, and use biochemical analyses to quantify the reactivity of inflammation, toxic as well as neurotrophic factors. Through the follow-up design, this study also plan to investigate the lasting duration of the intervention and the how the neural reorganization occurs as function of time.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 50 years old.
2. Diagnosed with subjective memory complaint (SMC) and with lower cognitive activities and physical activities.
3. Voluntary to sign the Informed Consent Form.

Exclusion Criteria:

1. Participants or first-degree relatives diagnosed with mental diseases.
2. Participants have history of severe neurological diseases or brain injury led to loss of consciousness.
3. Participants have diagnosis of cardiovascular disease.
4. Participants have History of alcohol, Nicotine, or substance dependence.
5. Participants suffer from visual, hearing degradation (including Hearing aid user).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in Electroencephalogram (EEG) performance. | baseline, post-treatment (6 months), follow-up (12 months)
  The amplitude, latency of MMN (mismatch negativity), N2, and the P3 components will be used to evaluate the memory and inhibitory control ability. Other EEG time-frequency analysis will be used to examine the changes of different frequency bands, such as theta, alpha, beta, and gamma.
Concentration change from baseline in the blood biochemical indices. (Total Tau, Aβ1-40, Aβ1-42, IL-1b, TNF-a, IL-6, TGF-b, BDNF, insulin, and ApoE4) | baseline, post-treatment (6 months), follow-up (12 months)
  Blood samples will use an enzyme-linked immunosorbent assay (ELISA) to assay the concentrations of Tau, Beta Amyloid (Aβ)1-40, Aβ1-42, interleukin-1β (IL-1β), tumor necrosis factor (TNF)-⍺, Interleukin-6 (IL-6), transforming growth factor (TGF)-β, brain-derived neurotrophic factor (BDNF), insulin, etc. The apolipoprotein E4 (ApoE4) genotype will also be evaluated.
Change score of the Chinese version Verbal Learning Test (CVVLT). | baseline, post-treatment (6 months), follow-up (12 months)
  A nine-item of CVVLT (total recall, delayed recall) will be applied to measure the participant's memory ability, with a higher score indicating better performance.
Change score of the WMS-III logical memory test part A. | baseline, post-treatment (6 months), follow-up (12 months)
  WMS-III logical memory test part A (immediate recall, delayed recall) will be applied to measure the participant's memory ability. The maximum score is 25 for each recall trial, with a higher score indicating better performance.
Change score of the Taylor Complex Figure Test (TCFT). | baseline, post-treatment (6 months), follow-up (12 months)
  TCFT (immediate recall, delayed recall) will be applied to measure the participant's memory ability. The maximum score is 36 for each recall trial, with a higher score indicating better performance.
Change score of the Digit Span Backward Test. | baseline, post-treatment (6 months), follow-up (12 months)
  The Digit Span Backwards Task will be applied to measure the participant's working memory ability. A higher score indicating better performance.

SECONDARY OUTCOMES:
Subjective memory complaint survey. | baseline, post-treatment (6 months), follow-up (12 months)
  A 14-item Subjective Memory Complaints Questionnaire measured memory impairment. The response was restricted to either "Yes" or "No".
Change scores of EuroQol-5 Dimension (EQ-5D). | baseline, post-treatment (6 months), follow-up (12 months)
  The EQ-5D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression to measure the quality of life. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Lifestyle activities survey. | baseline, post-treatment (6 months), follow-up (12 months)
  This self-report questionnaire measured the frequency of cognitive (e.g. read newspaper, go to museum) and physical activities (e.g.jogging, swimming). Each activity has four levels to rate frequency, with the lower score means a lower frequency on that activity.
Physiological parameter (Blood pressure and blood glucose) survey. | baseline, post-treatment (6 months), follow-up (12 months)
  The data will be used to evaluate whether lifestyle remodeling intervention regulates the values of the physiological parameters(blood pressure and blood glucose level), further to investigate the association between physiological parameters and cognitive function.
Change score of the Cognitive Abilities Screening Instrument (CASI). | baseline, post-treatment (6 months), follow-up (12 months)
  CASI will be applied to measure the participant's general cognitive ability. The range of score is 0 to 100, with a higher score indicating better performance.
Change score of the Boston Naming Test (BNT). | baseline, post-treatment (6 months), follow-up (12 months)
  Thirty-item version BNT will be applied to measure the participant's linguistic ability. The maximum score is 25, with a higher score indicating better performance.
Change score of the category Verbal Fluency Test (VFT). | baseline, post-treatment (6 months), follow-up (12 months)
  The category VFT will be applied to measure the participant's language and executive function, with a higher score indicates better performance.
Performance changes of the Trail Making Test Form A/B (TMT-A/B). | baseline, post-treatment (6 months), follow-up (12 months)
  TMT-A/B will be applied to measure participant's attention and executive function.
  The number of seconds to complete each trial and the number of errors would be recorded, with a higher value indicating greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ning Wang, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No